CLINICAL TRIAL: NCT00806481
Title: Does Phosphate Binding With Sevelamer Carbonate Improve Cardiovascular Structure and Function in Patients With Early Chronic Kidney Disease?
Brief Title: Effects of Phosphate Binding With Sevelamer in Stage 3 Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Charles Ferro, Dr, Consultant Nephrologist and Honorary Senior Lecturer, University Hospital Birmingham NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RRK3563; SVCARB01508IST; 2008-003727-23
Record Dates: First submitted 2008-06-25; First posted 2008-12-10 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Kidney Failure, Chronic; Cardiovascular Diseases
Keywords: Phosphate
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Treatment group: treatment with 1600mg tablets of sevelamer carbonate three times daily for 36 weeks
  Interventions: Drug: Sevelamer carbonate
- 2 (Placebo Comparator): Treatment group: treatment with tablets of placebo three times daily for 36 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sevelamer carbonate — Treatment group: treatment with 1600mg tablets of sevelamer carbonate three times daily for 36 weeks
  Other Names: Sevelamer carbonate (Renvela)
  Arms: 1
Drug: Placebo — Treatment group: treatment with tablets of placebo three times daily for 36 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether lowering phosphate in patients with early chronic kidney disease with the phosphate binder sevelamer has beneficial effects on cardiovascular structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients aged 18 to 80 years
* Chronic kidney disease stage 3 (defined as a glomerular filtration rate of 30-60 ml/min/1.73m2)
* Office blood pressure controlled to less than 140/90 mmHg for 12 months before entry into the study
* Total cholesterol less than 5.5 mmol/l

Exclusion Criteria:

* Existing or previous treatment within 1 year with a phosphate binder or vitamin D analogue
* Uncontrolled hyperphosphataemia (serum phosphate >1.8 mmol/l)
* Uncontrolled secondary hyperparathyroidism (PTH >80 pg/ml)
* Diabetes mellitus
* Pregnancy
* Moderate-severe cardiac valvular disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass | 36 weeks

SECONDARY OUTCOMES:
Aortic compliance as measured by cardiac magnetic resonance imaging | 36 weeks
Arterial stiffness as measured by pulse wave velocity and pulse wave analysis | 36 weeks
Arterial elastance as measured by echocardiography | 36 weeks
Left ventricular systolic and diastolic elastance measured by echocardiography | 36 weeks
Bone density on dual-energy x-ray absorptiometry scanning | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Ferro, BSc (Hons), MBChB, FRCP, MD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Chue CD, Townend JN, Steeds RP, Ferro CJ. Evaluating the effects of sevelamer carbonate on cardiovascular structure and function in chronic renal impairment in Birmingham: the CRIB-PHOS randomised controlled trial. Trials. 2011 Feb 2;12:30. doi: 10.1186/1745-6215-12-30. PMID 21288351